CLINICAL TRIAL: NCT07296315
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Confirm Efficacy and Safety of MH002 and to Assess the Effect of Dose in Patients With Mild-to- Moderate Ulcerative Colitis Insufficiently Controlled With 5-Aminosalicylic Acid
Brief Title: Confirmatory Clinical Study in Active Ulcerative Colitis
Acronym: StarFish-UC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MRM Health NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MH002-UC-202
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Colitis, Ulcerative
Keywords: 5-aminosalicylic-acid; live biotherapeutic product; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-dose MH002 (Experimental)
  Interventions: Drug: Low-dose MH002
- High-dose MH002 (Experimental)
  Interventions: Drug: High-dose MH002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose MH002 — Microbiome-based live biotherapeutic product consisting of 6 wildtype commensal strains at a dose of 1 × 10^10 equivalent colony forming units [eqCFU]), administered orally (in a capsule) once daily
  Arms: Low-dose MH002
Drug: High-dose MH002 — Microbiome-based live biotherapeutic product consisting of 6 wildtype commensal strains at a dose of 4 × 10^10 equivalent colony forming units [eqCFU]), administered orally (in a capsule) once daily
  Arms: High-dose MH002
Drug: Placebo — Blank placebo administered orally (in a capsule) once daily
  Arms: Placebo

SUMMARY:
The main goal of the study is to check if MH002 works and is safe to use. In a previous study in 45 patients with Ulcerative Colitis, MH002 was found to have favorable effects. In this study, 2 different doses will be tested, and long-term treatment effects will be investigated.

MH002 is a live biotherapeutic product (LBP). This is a biological medicine containing live bacteria used to restore the normal function of a gut that is damaged by ulcerative colitis (UC). Ulcerative colitis is a bowel disease that causes inflammation and sores in the gut.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis (histologic diagnosis and either endoscopic or radiographic diagnosis) of ulcerative colitis (UC) at least 3 months prior to Screening.
* Diagnosis of active mild-to-moderate UC at Screening as defined by an mMS of 4 to 7, including a MES ≥2 (confirmed by central reading), a Mayo Rectal Bleeding score of 1 or 2, and a Mayo Stool Frequency score ≥1.
* UC lesions extending ≥10 cm from the anal verge.
* Participant must either receive a stable dose of orally administered 5-aminosalicylic acid (5-ASA); have failed, due to insufficient efficacy, oral 5-ASA; have a documented intolerance or poor tolerance to an aminosalicylic acid treatment, including 5-ASA, or be contra-indicated to receive 5-ASA treatment per local labeling.
* Participant must provide written informed consent or assent (parent or legal guardian must provide consent for a participant <18 years of age who has assented to participate in the study, or as required per local regulations).
* In countries not allowing females of childbearing potential (FOCBP) to participate without an acceptable contraceptive method, the FOCBP must agree to abide to local requirements and eg, use at least an acceptable method of contraception until the end of treatment.

Exclusion Criteria:

* Diagnosis of Crohn's disease, undetermined colitis, ischemic colitis, fulminant colitis, or toxic megacolon.
* Evidence of a clinically significant, active infection of the gastrointestinal tract.
* Severe UC (mMS>7), meeting modified Truelove Witts' criteria and/or RB score of 3, participant with ulcerative proctitis only, or participant in whom colitis is most severe in the transverse colon or ascending colon, or if any hospitalization is planned at the time of Screening.
* Total colectomy, stoma, or ileo-anal pouch, or history of extensive colonic resection leaving less than 30 cm of colon.
* Presence of intra-abdominal fistula, abscesses, diverticulitis, or gastrointestinal bleeding unrelated to UC.
* History of colon carcinoma or high-grade dysplasia.
* Previous use of any advanced UC treatment, including any anti-TNF (eg, infliximab), antiintegrin (eg, vedolizumab) or anti-IL-12/23 (eg, ustekinumab) agent, anti-IL23 (eg, risankizumab), Janus kinase inhibitors (eg, tofacitinib), and sphingosine-1-phosphate receptor modulators (eg, etrasimod).
* Use of sulfasalazine ≤4 weeks prior to randomization.
* Use of corticosteroids or any disease-modifying antirheumatic drugs (DMARD), including thiopurines, ≤6 weeks prior to randomization into the study, except for a stable, low dose of oral corticosteroids (≤10 mg prednisolone/day) for at least 2 weeks prior to Screening colonoscopy and up to at least the Week 12 visit.
* Use of antibiotics (except for local use), prebiotics, or probiotics ≤4 weeks prior to randomization or anticipated during study participation, or concomitant, chronic use of an antidiarrheal drug, or concomitant use of any rectal treatment.
* Use of fecal microbiota transplantation (FMT) ≤52 weeks prior to randomization.
* Treatment with another investigational drug or intervention within 30 days prior to Screening, or within 5 times the elimination half-life of the investigational drug (whichever is longest).
* Any immunocompromised state, including conditions linked to severe immunosuppression (eg, active human immunodeficiency virus, malignancies, liver cirrhosis, systemic chemotherapy).
* Leukopenia (total white blood cell count <3000/μL) and/or neutropenia (absolute neutrophil count <1000/μL), anemia (hemoglobin <10.0 g/dL), thrombocytopenia (peripheral blood platelet count <100 × 10^9/L), and/or any coagulation disorder with significantly increased risk of bleeding.
* Ongoing or recent (<3 months) renal disease or insufficiency as manifested, eg, by medical history and/or clinical examination and/or (calculated or measured) glomerular filtration rate ≤60 mL/min.
* Ongoing or recent (<3 months) advanced hepatic dysfunction defined as a Child Pugh score ≥10 (Class C), or increase ≥2 times the upper limit of normal in aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT) or international normalised ratio (INR).
* Clinically significant bone marrow disease if progressive or not controlled, or any history of solid organ or bone marrow transplantation.
* Active intravenous drug abuse or alcohol abuse disorder as assessed by the Investigator.
* Pregnancy or lactation at study entry. Note: Participants who become pregnant or start to breastfeed during the study may continue the study per the Investigator's discretion.
* Participants who are inappropriate for the study per the Investigator's discretion.
* An employee (or a relative of) of the Investigator, study center, contract research organization, or Sponsor.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in centrally-assessed Mayo Endoscopic Subscore (MES) at Week 12 | Week 12

SECONDARY OUTCOMES:
To confirm the efficacy of MH002 to induce clinical remission at Week 12 | Week 12
  Key secondary endpoint: Clinical remission is defined as a modified Mayo Score (mMS) ≤2, all mMS subscores ≤1, and an Rectal Bleeding (RB) subscore of 0, with endoscopic MES based on worst segment assessed by a blinded central reader, and 2-item Patient-Reported Outcome (PRO-2) scores computed from the e-diary data
Change from baseline in histologic scores Robarts' Histopathology Index (RHI) at Week 12 | Week 12
(Median) Percent change from baseline in fecal calprotectin (FC) at Week 12 | Week 12
Change from baseline in UC-100 score at Week 12 | Week 12
Change from baseline in PRO-2 score at Week 12 | Week 12
  2-item Patient-Reported Outcome (PRO-2) scores computed from the e-diary data
To confirm the safety and tolerability of MH002 in the Induction Phase | Up to Week 12
  * TEAEs and SAEs
  * Treatment-emergent abnormalities in laboratory parameters and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Ludo Haazen, MD, Study Chair — MRM Health NV
Locations (1):
- Peters Medical Research, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No